CLINICAL TRIAL: NCT00001807
Title: (1)H-Nuclear Magnetic Resonance Spectroscopic Imaging of the Brain in Patients Who Receive Neurotoxic Therapy
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990088; 99-C-0088; NCT00020293 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04-18

CONDITIONS: Brain Cancer; Brain Neoplasms
Keywords: CNS directed therapy; Neurotoxicity; H-NMRS; MRI
MeSH Terms: conditions — Brain Neoplasms; Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Central nervous system toxicity is a recognized side effect of certain therapies for cancers, particularly cranial irradiation, intrathecal therapy or systemic high-dose chemotherapy. The pathophysiologic mechanisms and clinical manifestations vary. Previous studies defining MRI changes and correlating these with neurocognitive deficiencies have been inconsistent. Recent advances in brain imaging may help to better define neurotoxic effects. (1)H-NMRS is a noninvasive method of obtaining in vivo biochemical information from the brain. It has been used to study patients with CNS disorders, including neuronal disorders. In this study, (1)H-NMRS will be used to objectively characterize CNS toxicities in patients with cancer who are receiving potentially neurotoxic therapies. In addition, we will retrospectively evaluate patients with known or suspected neurotoxicity associated with cancer therapy, to determine if changes in spectroscopic patterns are associated with CNS toxicity.

DETAILED DESCRIPTION:
Background:

* Central nervous system toxicity is a recognized side effect of certain cancer therapies, particularly cranial irradiation, intrathecal therapy and systemic high-dose chemotherapy.
* The pathophysiologic mechanisms are not well-defined and clinical manifestations vary. Previous studies defining MRI changes and correlating these with neurocognitive deficiencies have been inconsistent.
* Recent advances in brain imaging may help to better define neurotoxic effects. (1)H-NMRS is a noninvasive method of obtaining in vivo biochemical information from the brain. It has been used to study patients with CNS disorders, including neuronal disorders.

Objective:

-To identify specific patterns of brain metabolites that are associated with therapy-related neurotoxicity using (1)H-NMRS in cancer patients who are receiving or have received potentially neurotoxic therapy.

Eligibility:

-Patients with brain tumors or patients receiving high-dose systemic chemotherapy, intrathecal chemotherapy (lumbar puncture or intra-Ommaya), or cranial radiation therapy OR patients with documented or suspected clinical neurotoxicity presumed to be caused by treatment for cancer.

Design:

* In order to identify metabolite profiles that may be associated with neurotoxicity, NMRS data will be collected in a cross-sectional manner from patients at various stages of treatment and longitudinally throughout the course of therapy.
* NMRS studies will be performed on patients entered on this study at any or all of the following times: prior to therapy, immediately after the first cycle of therapy, prior to subsequent cycles of therapy, or after completion of all therapy.
* Neurotoxicity will also be evaluated by neuropsychological testing.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with brain tumors or patients receiving high-dose systemic chemotherapy, intrathecal chemotherapy (lumbar puncture or intra-Ommaya), or cranial radiation therapy or patients with documented or suspected clinical neurotoxicity presumed to be caused by treatment for cancer.

Durable Power of Attorney (DPA) should be offered to all patients greater than or equal to 18 years of age.

All patients or their legal guardians (if the patient is less than 18 years of age) must sign a document of informed consent indicating their awareness of the investigational nature and the risks of this study. When appropriate, the minor patient will sign a written assent.

EXCLUSION CRITERIA:

Pregnancy.

Patients with braces or permanent retainers.

Patients with pre-existing neurologic or genetic conditions, unrelated to the tumor.

Patients who are unable (either because of physical or psychological factors) to undergo imaging studies and who are not a candidate for anesthesia.

Patients who have an absent gag reflex or swallowing difficulties.

Metallic implants, including cardiac pacemakers, neural pacemakers, shrapnel, cochlear implants or ferrous surgical clips.

History of severe reaction to Gadolinium.

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 1999-04-16; Study Completion 2019-04-18

PRIMARY OUTCOMES:
Identify patterns of brain metabolites associated with therapy related neurotoxicity | At time of MRI and till date of death
  changes in spectroscopic metabolite patterns defined by neuropsychological testing or abnormalities on conventional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brown RT, Madan-Swain A, Pais R, Lambert RG, Sexson S, Ragab A. Chemotherapy for acute lymphocytic leukemia: cognitive and academic sequelae. J Pediatr. 1992 Dec;121(6):885-9. doi: 10.1016/s0022-3476(05)80333-6. PMID 1447650
- [Background] Ochs J, Mulhern R, Fairclough D, Parvey L, Whitaker J, Ch'ien L, Mauer A, Simone J. Comparison of neuropsychologic functioning and clinical indicators of neurotoxicity in long-term survivors of childhood leukemia given cranial radiation or parenteral methotrexate: a prospective study. J Clin Oncol. 1991 Jan;9(1):145-51. doi: 10.1200/JCO.1991.9.1.145. PMID 1985164
- [Background] Hoppe-Hirsch E, Renier D, Lellouch-Tubiana A, Sainte-Rose C, Pierre-Kahn A, Hirsch JF. Medulloblastoma in childhood: progressive intellectual deterioration. Childs Nerv Syst. 1990 Mar;6(2):60-5. doi: 10.1007/BF00307922. PMID 2340529